CLINICAL TRIAL: NCT03910634
Title: IMRT Combined With Carboplatin Versus IMRT Combined With Carboplatin and Fluorouracil in the Treatment of Locally Advanced Esophageal Cancer in Elderly Patients With High Risk of Chemotherapy: a Randomized Controlled Clinical Study
Brief Title: IMRT With Carboplatin Versus IMRT With Carboplatin and Fluorouracil for Eldly Esophageal Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhu Yujia, Doctor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GD-Q201807
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Esophageal Cancer; Radiotherapy Side Effect
Keywords: Esophageal Cancer; radiotherapy; chemotherapy; Carboplatin
MeSH Terms: conditions — Esophageal Neoplasms; Radiation Injuries | interventions — Fluorouracil; Radiotherapy, Intensity-Modulated; Carboplatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMRT combined with carboplatin (Experimental): Intensity modulated radiation therapy 50-60Gy, Carboplatin (AUC 2), QW1, intravenous drip, repeat for 4 weeks
  Interventions: Radiation: Intensity modulated radiation therapy; Drug: carboplatin
- IMRT combined with carboplatin and fluorouracil (Placebo Comparator): Intensity modulated radiation therapy 50-60Gy, Carboplatin (AUC 2), QW1, intravenous drip; Fluorouracil 1.33g/body surface QW1, continuous intravenous infusion for 72 hours, repeated for 4 weeks
  Interventions: Drug: Fluorouracil; Radiation: Intensity modulated radiation therapy; Drug: carboplatin

INTERVENTIONS:
Drug: Fluorouracil — 1.33g/body surface QW1, continuous intravenous infusion for 72 hours, repeated for 4 weeks
  Other Names: 5-FU
  Arms: IMRT combined with carboplatin and fluorouracil
Radiation: Intensity modulated radiation therapy — Radiotherapy for 5-6 weeks，50-60Gy
  Other Names: IMRT
Drug: carboplatin — Carboplatin (AUC 2), QW1, intravenous drip, repeat for 4 weeks

SUMMARY:
An open, single-center, randomized controlled phase II clinical trial to compare the efficacy and safety of conformal intensity modulated radiation therapy (IMRT) combined with carboplatin and IMRT combined with carboplatin and 5-FU in elderly patients with locally advanced esophageal squamous cell carcinoma at high risk of chemotherapy

DETAILED DESCRIPTION:
Esophageal cancer is one of the most common malignant tumors in China.To compare the efficacy and safety of conformal intensity modulated radiation therapy (IMRT) combined with carboplatin and IMRT combined with carboplatin and 5-FU in elderly patients with locally advanced esophageal squamous cell carcinoma at high risk of chemotherapy.This trial is an open, single-center, randomized controlled phase II clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age (> 65 years)
* Histologically confirmed esophageal squamous cell carcinoma, the 8th edition of AJCC stage T3-4NxM0 or TxN1-3M0, without surgical indications after consultation by surgeons.
* PS score < 2, Chemotherapy risk score is medium and high risk
* No radical thoracic surgery/chemotherapy/radiotherapy/targeted therapy has been performed in the past.
* Diseases measurable according to RECIST standards
* Hematological examination requires Hb (>90g/L), ANC (>2.0 *109/L) and platelet (>100 *109/L). Serum albumin (>3.0g/dL)
* Serum creatinine < 1.25 times normal upper limit (UNL), or creatinine clearance rate (>60 ml/min). Total bilirubin < upper limit of normal value
* Total bilirubin < the upper limit of normal value, AST (SGOT) and ALT (SGPT) < 2.5 times the upper limit of normal value, ALP < 2.5 times the upper limit of normal value (ULN)
* If exploratory surgery is performed, the patient will recover at least 2 weeks after operation.

Exclusion Criteria:

* Pregnant or lactating women.
* Patients with fertility without adequate contraceptive measures.
* Anaphylaxis to 5FU and carboplatin is known.
* Anaphylaxis known to exist with any drug in the study
* Other malignant tumors have occurred in the past five years, except cervical carcinoma in situ or non-melanoma skin cancer, which has been properly treated.
* Discovery of esophageal fistula or risk of esophageal bleeding before treatment
* Distant organ metastasis is known
* Symptomatic peripheral neuropathy, according to NCIC-CTC criteria (> grade 2).
* Other serious diseases or medical conditions: Myocardial infarction (in the past six months), severe unstable angina pectoris and congestive heart failure have occurred.
* Severe complications (including intestinal paralysis, intestinal obstruction, interstitial pneumonia, pulmonary fibrosis, severe respiratory dysfunction of COPD, cardiac dysfunction of pulmonary heart disease, uncontrolled diabetes mellitus, renal insufficiency and cirrhosis of liver, etc.)
* Gastrointestinal bleeding requires frequent blood transfusion.
* It is known to carry human immunodeficiency virus (HIV) or AIDS.
* Suffering from mental illness
* The known neuropathy is of grade 2 or higher severity.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2019-04-09 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall objective response rate | up to 24 months
  The proportion of partial and complete remission of tumors

SECONDARY OUTCOMES:
Incidence of toxic and side effects above 3 degrees | up to 24 months
  The Incidence of toxic and side effects above 3 degrees in overall patients

CONTACTS AND LOCATIONS:
Overall Officials: Yonghong Hu, Doctor, Study Director — Sun Yat-sen University
Locations (1):
- SYSU Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No